CLINICAL TRIAL: NCT04251377
Title: Single-stage Surgery With Antibiotic-loaded Hydrogel Coated Implants Versus Two Stage Surgery for Secondary Prevention of Complex Chronic Periprosthetic Hip Joint Infection SINBIOSE-H.
Brief Title: Single-stage Surgery With Antibiotic-loaded Hydrogel Coated Implants Versus Two Stage Surgery for Secondary Prevention of Complex Chronic Periprosthetic Hip Joint Infection
Acronym: SINBIOSE-H
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18PH222; ANSM (Other: 2019-A01491-56)
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Hip Prosthesis Infection
Keywords: Surgery; Biofilm inhibitor; Chronic infections; Total Hip Arthroplasties (THA); Defensive Antibacterial Coating (DAC®); Novagenit®; Hip Prosthesis
MeSH Terms: conditions — Persistent Infection; Limb Deficiencies, Distal, with Micrognathia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-stage surgery + DAC® + topical antibiotics (Experimental): Experimental group is composed of single-stage procedure associated to the use of biofilm inhibitor (Defensive Antibacterial Coating® DAC®) and topical antibiotics=new strategy
  Interventions: Device: Defensive Antiadhesive Coating DAC®, Novagenit SRL
- control group : two-stage surgery (No Intervention): Control group is composed of two-stage procedure without biofilm inhibitor (standard protocol)

INTERVENTIONS:
Device: Defensive Antiadhesive Coating DAC®, Novagenit SRL — DAC gel, mixed with topical antibiotics is applied on the surface of the implants before implantation, in a sterile environment in the operating room.
  The topical antibiotics will be added to the reconstituted DAC® gel preparation, at the discretion of the physician, on the basis of pre-operative culture.
  Arms: Single-stage surgery + DAC® + topical antibiotics

SUMMARY:
Each year, around 1500 infected Total Hip Arthroplasties (THA) need non-conservative surgery, remaining an issue for patients and healthcare units. The recommended treatment, relying on cohort reviews and international consensus follows a two-stage protocol. This protocol implies a first surgery to remove all infected implants and at least 6 weeks of antibiotic treatment without implant, then usually an antibiotic-free period and only then a second surgery to put back new implants and start the rehabilitation protocol, with usually more than a week of a second hospital stay. Between both surgeries, full-weight bearing is prohibited and joint stiffness and/or pain are rather usual complications. Failure rate is estimated at 10% in this two-stage strategy. The single-stage procedure (i.e. implanting back a new prosthesis during the same surgery after implant removal, synovectomy and lavage) is thought to be less susceptible to late functional complications (i.e. pain, stiffness and muscle deficiency) with a shorter, single hospital stay.

Although, with single-stage surgery, infection control could be less efficient because most pathogens produce during the first hours of infection an antibiotic-resistant layer called biofilm, allowing them to colonize and adhere to foreign objects like implants. This single-surgery protocol thus highly relies on antibiotics and has a list of contra-indications (based on experts' consensus): the presence of damaged soft tissues or a sinus tract, unknown pathogens, difficult to treat micro-organisms, severe immunosuppression and for many surgeons, each time a bone graft is necessary. Most of these contra-indications are directly related to the biofilm.

As no randomized control trial has ever compared single-stage versus two-stage surgery, the level of evidence for recommending one procedure over the other is low.

We conducted a survey that showed that most of the French reference centers have already switched to single stage surgery for single-stage non contra-indicated cases.

An antibiotic-loaded hydrogel coating (Defensive Antiadhesive Coating®, Novagenit SRL), has been proven to mechanically prevent the biofilm formation, while allowing a prolonged intraarticular antibiotic release, in a randomized controlled trial in primary prevention of infection in THA.

The addition of this biofilm inhibitor to a single-stage surgery might stand as a promising strategy for secondary prevention of peri-prosthetic hip joint infection. Moreover, using this device to prevent biofilm formation could expand one stage surgery to patients that are "normally" contra-indicated to one stage surgery.

ELIGIBILITY:
Inclusion Criteria:

* Social security affiliation
* Signed informed consent
* Chronic periprosthetic hip joint infection defined according to the Musculoskeletal Infection Society criteria :
* Two positive periprosthetic cultures with phenotypically identical organisms
* or a sinus tract communicating with the joint,
* or having 3 of 5 minor criteria:

  * Elevated serum C-reactive protein (CRP) and Erythrocyte Sedimentation Rate (ESR);
  * Elevated synovial fluid White Blood Cell (WBC) count or change of ++ on leukocyte esterase test strip;
  * Elevated synovial fluid Polymorphonuclear Neutrophil Percentage (PMN%);
  * Positive histological analysis of periprosthetic tissue;
  * A single positive culture.

Exclusion Criteria:

* Patients with hypersensitivity to hydrogel components (hyaluronic acid and/or poly-lactic acid) known of Defensive Antibacterial Coating (DAC)®
* Pregnancy or positive pregnancy test (performed in women of childbearing age before inclusion)
* Life expectancy < 3 months
* Expected use of a cemented implant by the surgical team (for the treatment surgical protocol)
* Unable to give informed consent
* Patients under guardianship or curators
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of clinically diagnosed infection relapse of the periprosthetic joint | Years : 2
  The periprosthetic joint infection is defined according to the Musculoskeletal Infection Society criteria:
  * Two positive periprosthetic cultures with phenotypically identical organisms
  * or a sinus tract communicating with the joint,
  * or having 3 of 5 minor criteria:
    * Elevated serum C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR);
    * Elevated synovial fluid white blood cell (WBC) count;
    * Elevated synovial fluid polymorphonuclear neutrophil percentage (PMN%);
    * Positive histological analysis of periprosthetic tissue;
    * A single positive culture.

SECONDARY OUTCOMES:
Harris Hip Score (HHS) results | Years : 2
  Harris Hip Score (HHS) contains 10 items with maximum score at 100 for a perfect hip and minimum score at 0 for a very bad result.
Postel-Merle d'Aubigné (PMA) results | Years : 2
  Postel-Merle d'Aubigné (PMA) contains 3 items (pain, mobility and functional hip) with maximum score at 18 for a perfect hip and minimum score at 0 for a very bad result.
Hip dysfunction and Osteoarthritis Outcome Score (HOOS) results | Years : 2
  Hip dysfunction and Osteoarthritis Outcome Score contains 6 items (symptoms, stiffness, pain, function and daily life, sport and leisure activities, quality of life) and measure everyday activities with score from 0 to 4.
Oxford-12 results | Years : 2
  Oxford-12 allows to know the feelings of the patient during the last 4 weeks felt from 1 to 5 (satisfaction score).
Death rate (%) | Years : 2
  Analysis of death rate by group.
Post-operative complications | Years : 2
  Analysis of post-operative complications by group.
Revision surgery for any cause other than infection | Years : 2
  Analysis of revision surgery for any cause other than infection.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand BOYER, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (14):
- France (14):
  - CHU Amiens, Amiens
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Lille, Lille
  - HCL - Hôpital de la Croix Rousse, Lyon
  - HCL - Hôpital Edouard Herriot, Lyon
  - CHU Marseille, Marseille
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Chu Saint-Etienne, Saint-Etienne
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boyer B, Cazorla C, Carricajo A, Labruyere C, Chapelle C, Presles E, Zufferey P, Botelho-Nevers E. Single-stage surgery with antibiotic-loaded hydrogel-coated implants versus two-stage surgery for chronic periprosthetic hip joint infection in French tertiary referral hospitals: the SINBIOSE-H non-inferiority, randomised, controlled trial study protocol. BMJ Open. 2025 Feb 25;15(2):e085146. doi: 10.1136/bmjopen-2024-085146. PMID 40000087